CLINICAL TRIAL: NCT02393885
Title: Pivotal Study Of A Dual Epicardial & Endocardial Procedure (DEEP) Approach for Treatment of Subjects With Persistent or Long Standing Persistent Atrial Fibrillation With Radiofrequency Ablation
Brief Title: Pivotal Study Of A Dual Epicardial & Endocardial Procedure (DEEP) Approach
Acronym: DEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AtriCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP2014-1
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Results first posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation; Persistent or Longstanding Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes

ARMS (1):
- AtriCure Bipolar System and AtriClip® PRO LAA Exclusion System (Experimental): AtriCure Bipolar System and AtriClip® PRO LAA Exclusion System at day 1 of surgical procedure followed by endocardial catheter ablation procedure to occur at approximately 90 days after day 1 of surgical procedure.
  Interventions: Device: AtriCure Bipolar System and AtriClip® PRO LAA Exclusion System, Endocardial Ablation

INTERVENTIONS:
Device: AtriCure Bipolar System and AtriClip® PRO LAA Exclusion System, Endocardial Ablation
  Other Names: Irrigated Endocardial Catheters

SUMMARY:
The objective of this study is to establish the safety and effectiveness of a dual epicardial and endocardial ablation procedure for patients presenting with Persistent Atrial Fibrillation or Longstanding Persistent Atrial Fibrillation

DETAILED DESCRIPTION:
The objective of this study is to establish the safety and effectiveness of a dual epicardial and endocardial ablation procedure for patients presenting with Persistent Atrial Fibrillation or Longstanding Persistent Atrial Fibrillation utilizing the AtriCure Bipolar System and AtriClip® PRO LAA Exclusion System in an endoscopic or open ablation procedure, followed by an endocardial mapping and ablation procedure utilizing commercially available RF based, irrigated, power controlled, ablation catheters for endocardial lesions. The endocardial procedure will be staged to occur after 90 days post epicardial surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic Persistent Atrial Fibrillation or Longstanding Persistent Atrial Fibrillation refractory to a minimum of one Class I or Class III AADs.

Exclusion Criteria:

1. AF >10 years.
2. Refractory hypertension, defined as systolic (>150 mm Hg) or diastolic (> 90 mm Hg) blood pressure that remains uncontrolled despite sustained therapy
3. History of pulmonary hypertension
4. Pulmonary vein stenosis in one or more of the pulmonary veins
5. EP catheter ablation procedure to treat atrial fibrillation within 3 months
6. Undergone prior cardiothoracic surgery, previous thorax trauma which resulted in a pneumothorax or hemothorax.
7. Sleep apnea, home oxygen therapy, moderate to severe COPD, (FEV1/FVC < 70% predicted) or patient is considered intolerant to single lung ventilation.
8. NYHA Class IV heart failure.
9. Uncorrected, reversible cause(s) of atrial fibrillation, or is currently being treated for arrhythmias other than atrial fibrillation (AF) or atrial flutter.
10. Documented history of previous catheter ablation with perforation, history of pericarditis, pericardial effusion, or tamponade.
11. Structural heart disease requiring surgical treatment (i.e. valve disease requiring repair or replacement within 12 months following surgical ablation procedure).
12. CAD requiring intervention (either surgical, i.e. CABG, or catheter).
13. Ejection fraction < 30%
14. Measured left atrial diameter > 5.5 cm
15. Stroke/cerebrovascular accident (CVA) within previous six months, carotid artery stenosis greater than 80%.
16. BMI is >40
17. Thrombus in the left atrium or the left atrial appendage, determined by echocardiography (either at baseline TTE (or equivalent diagnostic test) or intraoperative TEE).
18. Blood dyscrasia or clotting disorder (i.e. Idiopathic Thrombocytopenic Purpura [ITP] or Thrombotic Thrombocytopenic Purpura [TTP]).
19. Contraindication to anticoagulation that in the opinion of the investigator poses undue risk to the patient from participating in the endocardial EP procedure.
20. Documented thromboembolism within the previous six months prior to signing informed consent.
21. Has the following atrial myxoma, mural thrombus or mural tumor.
22. A condition or congenital anomaly which prevents required surgical or catheter access.
23. A co-morbid condition that, in the opinion of the investigator, poses undue risk of general anesthesia or port access cardiac surgery.
24. Currently abusing drugs or alcohol.
25. Currently or has participated in a clinical study in the last 3 months prior to signing informed consent.
26. A psychological disorder that could interfere with provision of informed consent, completion of tests, therapy, or follow-up.
27. A condition that, in the opinion of the investigator, may jeopardize the patient's well-being and/or the soundness of this clinical study.
28. Pre-existing esophageal condition that required (or requires) endoscopic therapy or surgical treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2024-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Ellenbogen, MD, Principal Investigator — VCU; Vigneshwar Kasirajan, MD, Principal Investigator — VCU; Ali Khoynezhad, MD, Principal Investigator — MemorialCare Long Beach Medical Ctr
Locations (17):
- United States (15):
  - Long Beach Memorial Medical Center, Long Beach, California
  - Cedars-Sinai Heart Institute, Los Angeles, California
  - Alta Bates Sutter Medical Center, East Bay Hospital, Oakland, California
  - St. Helena Hospital, Adventist Heart Institute, St. Helena, California
  - Stanford University Department of CV medicine, Stanford, California
  - Shands at the University of Florida, Gainesville, Florida
  - Orlando Heart Institute, Orlando, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - The Christ Hospital, Cincinnati, Ohio
  - Tri Health Hosptial - Good Samaritan and Bethesda North Hospitals, Cincinnati, Ohio
  - Pinnacle Health, Harrisburg, Pennsylvania
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Aspirus Research Institute, Wausau, Wisconsin
- Universitair Ziekenhuis Brussel (UZ Brussels), Brussels, Belgium
- Academic Medical Center (AMC), Amsterdam, Netherlands

REFERENCES:
- [Derived] Ellenbogen KA, Khoynezhad A, La Meir M, de Asmundis C, Koneru JN, Johnkoski J, Rist K, Mumtaz M, Link MG, de Groot JR, Driessen AHG, Lee MY, Hoff SJ, Bello D, Dunnington G, Eisenberg S, Vloka M, Taylor BJ, Jones SD, Philpott JM, Beaver TM, Miles WM, Khan JH, Kang S, Gandhi GD, Okum EJ, Badhwar N, Baykaner T, Lee AM, Vesco PA, Smith JM, Gaynor S, Frazier K, Lee RJ, Kasirajan V. Dual Epicardial and Endocardial Procedure (DEEP) for Persistent or Longstanding Persistent Atrial Fibrillation. Circ Arrhythm Electrophysiol. 2025 Oct;18(10):e013692. doi: 10.1161/CIRCEP.125.013692. Epub 2025 Sep 30. PMID 41025224

RESULTS

PARTICIPANT FLOW:
Groups:
- AtriCure Bipolar System and AtriClip® PRO LAA Exclusion System: AtriCure Bipolar System and AtriClip® PRO LAA Exclusion System at day 1 of surgical procedure followed by endocardial catheter ablation procedure to occur at approximately 90 days after day 1 of surgical procedure.
  AtriCure Bipolar System and AtriClip® PRO LAA Exclusion System, Endocardial Ablation
Period: Overall Study
Arm/Group | AtriCure Bipolar System and AtriClip® PRO LAA Exclusion System
Started | 90
Completed | 85
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | AtriCure Bipolar System and AtriClip® PRO LAA Exclusion System
Number analyzed (Participants) | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 48
  >=65 years | 42
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 90
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 87
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  Netherlands | 7
  Belgium | 14
  United States | 69

OUTCOME MEASURES:

1. Primary Outcome: Primary Effectiveness Endpoint
Description: Freedom from any documented AF, atrial flutter, or atrial tachycardia lasting >30 seconds in duration through the 12 month follow-up visit in the absence of Class I or III AADs (with the exception of previously failed AADs at doses not exceeding those previously failed).
Time Frame: 6 months post the Endocaridal Ablation Procedure through the 12 month follow-up visit
Population: Modified Intent to Treat (mITT)
Measure: Count of Participants; unit: Participants
Arm/Group | AtriCure Bipolar System and AtriClip® PRO LAA Exclusion System
Number analyzed (Participants) | 85
Participants | 61

2. Primary Outcome: Primary Safety Endpoint
Description: The primary safety endpoint is a composite endpoint consisting of any one or more of the events if they were adjudicated by the CEC to be serious adverse events (SAEs) and related to device/procedures as follows:
  1. The AtriCure Bipolar System and/or the AtriClip Pro LAA Exclusion System, within 30 days following the epicardial surgical ablation procedure; or
  2. The epicardial surgical ablation procedure within 30 days following the epicardial procedure; or
  3. The endocardial index procedure (or a repeat endocardial ablation procedure performed during the blanking period) within 7 days following an endocardial ablation procedure.
Time Frame: 30 Days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | AtriCure Bipolar System and AtriClip® PRO LAA Exclusion System
Number analyzed (Participants) | 90
Participants | 6

ADVERSE EVENTS:
Time Frame: 24 months
Description: All adverse events that occurred within 24 months post procedure were collected
Arm/Group | AtriCure Bipolar System and AtriClip® PRO LAA Exclusion System
All-Cause Mortality (participants affected / at risk) | 1/90
Serious Adverse Events (participants affected / at risk) | 24/90
Other Adverse Events (participants affected / at risk) | 23/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AtriCure Bipolar System and AtriClip® PRO LAA Exclusion System (N=90)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 3 (4)
Atrial tachycardia (Cardiac disorders) | 2 (3)
Atrioventricular block (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1)
Bursitis infective (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Pneumococcal sepsis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Atrio-oesophageal fistula (Injury, poisoning and procedural complications) | 1 (1)
Diaphragmatic injury (Injury, poisoning and procedural complications) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal haematoma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Air embolism (Vascular disorders) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1)
Femoral artery aneurysm (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AtriCure Bipolar System and AtriClip® PRO LAA Exclusion System (N=90)
Pericarditis (Cardiac disorders) | 5 (5)
Chest pain (General disorders) | 3 (3)
Oedema peripheral (General disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypertension (Vascular disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/85/NCT02393885/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/85/NCT02393885/SAP_001.pdf